CLINICAL TRIAL: NCT04432610
Title: Echocardiographic Study of a Single Dose Bisoprolol Versus Nebivolol in Healthy Subjects: a Randomized, Double-blind, Cross-over Study
Brief Title: Echocardiographic Study of a Single Dose Bisoprolol Versus Nebivolol in Healthy Subjects
Acronym: BINEB
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID pandemic
Sponsor: Clinical Hospital Center Zemun (Other)
Responsible Party: Principal Investigator, Ivan Stankovic, Head of Echocardiography, Clinical Hospital Center Zemun
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 01-2020
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Bisoprolol Adverse Reaction; Nebivolol Adverse Reaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bisoprolol first, Nebivolol Second (Experimental): In this arm, patient will first receive bisoprolol, and after 1 week washout period, nebivolol
  Interventions: Drug: Bisoprolol versus Nebivolol
- Nebivolol first, Bisoprolol second (Experimental): In this arm, patient will first receive nebivolol, and after 1 week washout period, bisoprolol
  Interventions: Drug: Bisoprolol versus Nebivolol

INTERVENTIONS:
Drug: Bisoprolol versus Nebivolol — All subjects will receive both drugs, but at different time periods determined by randomization, with 1 week washout period

SUMMARY:
This is a randomized, double-blind, crossover study in healthy adult subjects. Each subject will receive a single dose of bisoprolol 5 mg p.o. and nebivolol 5 mg p.o. with 1 week washout period. All subjects will undergo a physical examination, 12-lead electrocardiography and a comprehensive echocardiographic study before the administration of the study drug and 5 hours thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects (male and female)
2. Age interval: 20-60 years old (inclusive)

Exclusion Criteria:

1. Any known absolute or relative contraindication to beta-blocker therapy
2. Poor echogenicity
3. A resting heart rate <60 bpm
4. A resting blood pressure < 110/70 mmHg

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2030-01 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Relative change (%) of cardiac output (CO) | Pre- and 5 hours post study drug administration
  CO (l/min), will be assessed by calculating stroke volume using pulsed-wave doppler (velocity time integral)

SECONDARY OUTCOMES:
Absolute and relative changes of left ventricular ejection fraction (%) | Pre- and 5 hours post study drug administration
  Ejection fraction will be measured using modified Simpson rule
Absolute and relative changes of global longitudinal strain (%) | Pre- and 5 hours post study drug administration
  Global longitudinal strain will be assessed using speckle tracking echocardiography
Absolute and relative changes of myocardial work (%) | Pre- and 5 hours post study drug administration
  Myocardial work will be assessed by using a dedicated commercially available software (GE, Norway)
Absolute and relative changes of atrial function (ml) | Pre- and 5 hours post study drug administration
  Atrial function will be assessed by measuring phasic volume changes during diastole
Absolute change of myocardial dispersion (ms) | Pre- and 5 hours post study drug administration
  Myocardial dispersion will be assessed by using speckle tracking echocardiography
Absolute and relative changes of TAPSE (tricuspid annular plane systolic excursion, mm) | Pre- and 5 hours post study drug administration
  TAPSE will be assessed by M-mode echocardiography
Absolute and relative changes of blood pressure (mmHg) | Pre- and 5 hours post study drug administration
  Brachial blood pressure will be measured by sphygmomanometer
Absolute and relative changes in atrial strain (%) | Pre- and 5 hours post study drug administration
  Atrial strain will be assessed using speckle tracking echocardiography
Absolute and relative changes of electrical dispersion (ms) | Pre- and 5 hours post study drug administration
  Electrical dispersion will be assessed by using 12-lead electrocardiogram
Absolute and relative changes of right ventricular fractional area change (%) | Pre- and 5 hours post study drug administration
  The parameter will be assessed by two-dimensional echocardiography
Absolute and relative changes of heart rate (bpm) | Pre- and 5 hours post study drug administration
  Heart rate will be measured by 12-lead electrocardiography
Absolute and relative changes of left ventricular twist (%) | Pre- and 5 hours post study drug administration
  Twist will be assessed by speckle tracking echocardiography
Absolute and relative changes of QTc interval (ms) | Pre- and 5 hours post study drug administration
  QTc interval will be measured by using 12-lead electrocardiography
Absolute and relative changes of mitral E/A ratio (%) | Pre- and 5 hours post study drug administration
  E/A ratio will be assessed by pulsed-wave Doppler
Absolute and relative change of mitral E/e prime ratio (%) | Pre- and 5 hours post study drug administration
  E/e prime ratio will be assessed by pulsed-wave and tissue Doppler echocardiography
Absolute and relative change of mitral E-wave deceleration time (ms) | Pre- and 5 hours post study drug administration
  E-wave deceleration time will be measured by pulsed-wave Doppler echocardiography
Absolute and relative changes of right ventricular global longitudinal strain (%) | Pre- and 5 hours post study drug administration
  Global strain will be assessed by using speckle tracking echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Centre Zemun, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No